CLINICAL TRIAL: NCT03650972
Title: Implementation of AFL Monitoring in Clinical (Lapsiveden Laktaattipitoisuuden Merkitys kliinisessä käytössä)
Brief Title: Implementation of AFL Monitoring in Clinical Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Susanna Koski, Medical Doctor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: T194/2018
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Labour Dystocia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A, Non-bicarbonate (No Intervention): When labour arrest is diagnosed and the first AFL > 12 mmol/L the participants will be randomized to two groups. In group A the labour is treated according to the hospital's current guidelines during labour arrest, i.e. the stimulation with oxytocin is started and AFL is measured again after one hour
- B, Bicarbonate group (Active Comparator): When labour arrest is diagnosed and the first AFL > 12 mmol/L the participants will be randomized to two groups. In group B the participant will drink bicarbonate (2 packages of Samarin®) dissolved in 200 ml of water. Then after one hour the AFL will be measured again and the stimulation with oxytocin will be started if there is no progress in the cervix.
  Interventions: Other: Samarin

INTERVENTIONS:
Other: Samarin — Arm: Active Comparator: B, Bicarbonate group When labour arrest is diagnosed and the first AFL > 12 mmol/L the participants will be randomized to two groups. In group B the participant will drink bicarbonate (2 packages of Samarin®) dissolved in 200 ml of water. Then after one hour the AFL will be measured again and the stimulation with oxytocin will be started if there is no progress in the cervix.
  Arms: B, Bicarbonate group

SUMMARY:
The overall objective of this randomized controlled trial is to develop a clinical standard procedure for measuring lactate in amniotic fluid (amniotic fluid lactate = = AFL) during childbirth before oxytocin stimulation is started. The aim is to reduce the need for emergency caesarean section during dysfunctional labour. The aim is also to study how different substances (oxytocin and Samarin®) affect uterine metabolic status during labour.

Labour dystocia, i.e. prolonged labour, occurs in up to 30% in primipara deliveries and in about 20% of all the deliveries. In 2016, in Finland oxytocin stimulation was used in 42% of all the deliveries.

The uterus, myometrium, is one of the largest muscles in the human body and consists mainly of smooth muscle cells. During the contractions the myometrial vessels also contract, causing momentary hypoxia and activation of anaerobic metabolism: O2 and pH levels of the muscle cell decreases and the lactate concentration increases. After the contraction, the blood circulation is restored and the anaerobic metabolites gradually dissolve. Myometrium requires a sufficiently long break between the contractions to recover. In dysfunctional labour the anaerobic metabolites accumulate in the myometrium. Accumulation of lactate has proved significantly to reduce the spontaneous contractions of myometrium and hinder myometrium calcium metabolism, which in turn reduces the strength of the contractions. Amniotic fluid lactate is known to reflect the metabolic state of the uterus during the labour.

Prolonged labour can in many aspects be compared to the athlete's tired muscles. Many of today's athletes try to control the accumulation of lactic acid in their muscles during training by drinking baking soda (bicarbonate) dissolved in water one hour before their physical activity. Bicarbonate is known to function as a lactic acid buffer. Bicarbonate is considered as food and is sold in grocery stores as baking soda and for example as Samarin®. Samarin® is safe to use during pregnancy because as a bicarbonate it does not pass through placenta and does not affect the fetus.

The trial aims to research if high AFL values (AFL > 12 mmol/L) in women with labour arrest are best treated by:

A) treating the labour according to the hospital's current guidelines during labour arrest, i.e. starting the stimulation with oxytocin and measuring the AFL again after one hour B) administering bicarbonate (Samarin®) dissolved in water one hour before starting the stimulation with oxytocin

ELIGIBILITY:
Inclusion Criteria:

* gestational age at least 37 + 0 weeks
* singleton pregnancy
* cephalic presentation
* active labor (regular painful contractions, effaced cervix open at least 3cm)
* arrested labour progress according partogram and clinic guidelines

Exclusion Criteria:

* intra uterine fetal growth retardation (> 22%)
* intra uterine fetal death
* threat of fetal asphyxia
* severe vaginal bleeding
* disproportion between the fetal head and the mother's pelvis
* hypertonic contractions (more than 5 in 10 minutes)
* known allergy or hypersensitivity to oxytocin or to any of derivatives
* women who cannot understand the information of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Spontaneus Vaginal delivery | by the end of the delivery

IPD SHARING:
Plan to Share IPD: No